CLINICAL TRIAL: NCT00144053
Title: A Phase Ⅲ Randomized Study of Mitomycin/Vindesine/Cisplatin Versus Irinotecan/Carboplatin Versus Paclitaxel/Carboplatin With Concurrent Thoracic Radiotherapy for Unresectable Stage Ⅲ Non-Small-Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: West Japan Thoracic Oncology Group (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WJTOG0105
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2006-01-06 (Estimated); Status verified 2005-08

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — CP protocol

INTERVENTIONS:
Drug: Cisplatin+Vindesine+MMC/ concurrent radiation
Drug: Irinotecan+Carboplatin/concurrent radiation
Drug: Paclitaxel+Carboplatin/concurrent radiation

SUMMARY:
To evaluate whether two weekly concurrent chemoradiotherapy regimens offer any advantage over concurrent chemoradiotherapy regimens with Cisplatin, Vindesine, Mitomycin for unresectable stage III NSCLC.

ELIGIBILITY:
Inclusion Criteria:

All patients had histologically or cytologically confirmed locally advanced NSCLC. All patients must not have undergone any previous therapy for NSCLC. Patients had to have measurable disease, an Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1, and to be less than 75 years old. Adequate organ (bone marrow, renal, liver, heart, and lung) function was required. All patients gave written informed consent.

Exclusion Criteria:

The exclusion criteria consisted of pulmonary fibrosis, pleural effusion, pregnancy, lactation, active concurrent malignancies, severe drug allergies, myocardial infarction, severe heart disease, uncontrollable diabetes mellitus, and infection. -

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450
Dates: Start 2001-04

PRIMARY OUTCOMES:
Survival

SECONDARY OUTCOMES:
safety

CONTACTS AND LOCATIONS:
Overall Officials: Hisao Uejima, MD, Principal Investigator — West Japan Thoracic Oncology Group

REFERENCES:
- See also: Related Info — http://www.wjtog.org/